CLINICAL TRIAL: NCT02217423
Title: The Relationship Between Abdominal Circumference and Cardiorespiratory Repercussions in Hospitalized Patients Submitted to Physical Therapy
Brief Title: Abdominal Circumference and Cardiorespiratory Repercussions in Patients Submitted to Physical Therapy
Acronym: RACCRPPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Bruno Martinelli, Me, Universidade Federal de Sao Carlos
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 34609514100005502
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Obesity, Abdominal; Lung Disease
Keywords: Physical Therapy Modalities; Respiration Disorders; Respiratory Therapy
MeSH Terms: conditions — Obesity, Abdominal; Lung Diseases; Respiration Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Obstructive increased AC (Experimental): Patient with obstructive respiratory disease with increased abdominal circumference.
  chest physiotherapy. Chest physiotherapy airway clearance modality. The protocol consisted of breathing exercises during 30 minutes and included: passive and localized exercises, deep diaphragmatic breathing and exercises on the chest wall (compression, vibration) and cough.
  Interventions: Other: Chest physiotherapy airway clearance modality
- Obstructive disfunction with normal AC (Experimental): Patients with obstructive respiratory disease with normal abdominal circumference.
  Patient with obstructive respiratory disease with increased abdominal circumference.
  chest physiotherapy. Chest physiotherapy airway clearance modality. The protocol consisted of breathing exercises during 30 minutes: passive and localized exercises, deep diaphragmatic breathing and exercises on the chest wall (compression, vibration) and cough.
  Interventions: Other: Chest physiotherapy airway clearance modality
- Restrictive increased AC (Experimental): Patients with restrictive respiratory disease with increased abdominal circumference. chest physiotherapy chest wall expansion.
  The protocol consisted of breathing exercises during 30 minutes: passive and localized exercises, deep diaphragmatic breathing and exercises of chest wall expansion (decompression) and incentive spirometry.
  Interventions: Other: Chest physiotherapy chest wall expansion
- Restrictive disfunction with normal AC (Experimental): Patients with restrictive respiratory disease with normal abdominal circumference.
  Chest physiotherapy chest wall expansion. The protocol consisted of breathing exercises during 30 minutes: passive and localized exercises, deep diaphragmatic breathing and exercises of chest wall expansion (decompression) and incentive spirometry.
  Interventions: Other: Chest physiotherapy chest wall expansion

INTERVENTIONS:
Other: Chest physiotherapy chest wall expansion — chest physiotherapy The protocol consisted of breathing exercises during 30 minutes: passive and localized exercises, deep diaphragmatic breathing and exercises of chest wall expansion (decompression, Incentive Spirometry).
  Other Names: Chest physiotherapy
  Arms: Restrictive disfunction with normal AC; Restrictive increased AC
Other: Chest physiotherapy airway clearance modality — The protocol will be consisted the breathing exercises during 30 minutes: passive and localized exercises, deep diaphragmatic breathing and exercises on the chest (vibration, compression) and active cough.
  Other Names: Chest physical therapy
  Arms: Obstructive disfunction with normal AC; Obstructive increased AC

SUMMARY:
The purpose of this study is to determine whether the hospitalized patients with increased waist circumference exhibit cardiorespiratory alterations after chest physical therapy.

DETAILED DESCRIPTION:
The physiotherapist assessment will consist of anthropometry (body mass index, abdominal circumference, adipometer); chest inspection and palpation, vital signs (blood pressure, heart rate, respiratory frequence, oxymetry), dyspnea index and capillar blood glucose; and later with pulmonary tests (thoracoabdominal perimetry, respiratory muscle strength and pulmonary volume and capacity). This will be a quasi-experimental study. Patients will be divided into four groups according to waist circumference (increased or not, with respect to cardiovascular risk) and respiratory disorders (obstructive and restrictive). After this assessment, chest physical therapy will begin according to the protocol for obstructive and restrictive respiratory disorders. The treatment will have an average duration of 30 minutes. At the end of treatment (single session) the patient will be assessed again after five and thirty minutes.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (> 18 years old), clinical stability characterized by axillary body temperature below 38 ° C, hemoglobin higher than 7 g / dL, oxygen saturation by pulse oximetry greater than or equal to 88%, mean arterial pressure (MAP) greater than 70 or less than 120 mm Hg, heart rate between 50 bpm to 140 bpm ; ability to understand, carry out the commands appropriately for evaluative tests, with the Glasgow Coma Scale score greater than 8, locomotor integrity of the lower limbs, spontaneous breathing, lack of hospital physiotherapy during hospitalization, prescription for respiratory therapy; bronchodilator, if applicable four hours before intervention.

Exclusion Criteria:

* inadequate perform to the maneuvers of the evaluation (e.g. spirometry), hemodynamic instability, thoracic dermal injury, disabling orthopedic complications that compromise the techniques of assessment and intervention, lymphedema of the trunk; sudden weight gain with edema in limbs, ascites, nephrotic syndrome, congestive heart failure, liver cirrhosis, erysipelas, deep vein thrombosis, heart bypass, heart transplantation, arrhythmias, atrioventricular block, severe dyspnea (Borg> 5), spinal cord injury, hemoptysis, osteoporosis, recent surgeries, coagulopathy, bronchopleural fistula, subcutaneous emphysema, presence of diabetes mellitus associated with cardiac autonomic dysfunction, bronchoconstriction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in spirometric measures. | Baseline, five and thirty minutes.
  The spirometry is used to assess chest volume and capacity of individual patients respiratory disease and their response to therapy and is regarded as the gold standard measure of respiratory function. The following variables were recorded; forced vital capacity, forced expiratory volume achieved in 1 second.

SECONDARY OUTCOMES:
Comparison of pulse oxymetry before/after chest physiotherapy. Comparison of blood pressure before/after chest physiotherapy. | Baseline, five and thirty minutes.
  The pulse oxymetry or pulse oximeter is used to measure peripheral oxygen saturation.
  The arterial blood pressure (systolic and diastolic) will be measured by sphygmomanometer to follow the displacement.

OTHER OUTCOMES:
Comparison of heart rate variability before/after chest physiotherapy. Comparison of thoracoabdominal perimetry before/after chest physiotherapy. | Baseline, five and thirty minutes.
  Heart rate variability has become the conventionally accepted term to describe variations of both instantaneous heart rate and intervals (time domain).
  Thoracoabdominal perimetry consists of a set of measurements of thoracic and abdominal circumferences during respiratory movements, and it aims at quantifying the thoracoabdominal mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Martinelli, Me, Principal Investigator — UFSCar
Locations (1):
- Hospital Estadual Manoel de Abreu, Bauru, São Paulo, Brazil